CLINICAL TRIAL: NCT02857803
Title: The Impact of Using an Interactive System, a Paper and Pencil Program or Conventional Methodologies in the Rehabilitation of Stroke Patients: a Randomised Controlled Trial
Brief Title: A Randomised Controlled Trial Comparing the Impact of Virtual Reality, Paper and Pencil and Conventional Methods on Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Serviço de Saúde da Região Autónoma da Madeira (SESARAM), E.P.E. (Unknown)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Professor Auxiliar, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 303891
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: Virtual Reality; Cognitive Rehabilitation; Motor Rehabilitation; Ecological validity; Personalisation
MeSH Terms: conditions — Stroke | interventions — Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Virtual Reality (Experimental): The Virtual Reality group will perform personalised activities of daily living in the context of a simulated city (Reh@City). The interaction with the virtual environment will be through a natural user interface.
  Interventions: Procedure: Virtual Reality
- Paper and Pencil (Active Comparator): The paper and pencil group will perform a set of cognitive paper and pencil tasks personalised to their deficits and generated automatically through a Task Generator.
  Interventions: Procedure: Paper and Pencil
- Conventional Therapy (Active Comparator): The Conventional Therapy group will perform the activities offered by the public health system, which are motor-focused.
  Interventions: Procedure: Conventional Therapy

INTERVENTIONS:
Procedure: Virtual Reality — Intervention of 30 minutes, 3 times a week until reaching 12 sessions.
  Arms: Virtual Reality
Procedure: Paper and Pencil — Intervention of 30 minutes, 3 times a week until reaching 12 sessions.
  Arms: Paper and Pencil
Procedure: Conventional Therapy — Intervention of 30 minutes, 3 times a week until reaching 12 sessions.
  Arms: Conventional Therapy

SUMMARY:
Virtual Reality allows the integration of both cognitive and motor rehabilitation in a more ecologically valid context. The purpose of this study is to determine whether this methodology has more impact on stroke rehabilitation than a paper and pencil personalised program and conventional therapy, which is motor-focused.

DETAILED DESCRIPTION:
Cognitive impairments after stroke are not always given sufficient attention despite its limitations in activities-of-daily- living (ADL's). Current cognitive rehabilitation methods mostly rely on paper-and-pencil tasks targeting isolated domains, which is not consistent with everyday-life. Besides limited ecological-validity, paper-and-pencil tasks are not accessible for most stroke patients whose dominant arm is paretic. Virtual Reality (VR) has shown to be a solution for the development of accessible and ecologically valid systems, but, does it have more impact than a paper and pencil personalised intervention?

Through a participatory design approach, with health professionals, the investigators have developed:

* a motor-accessible and cognitive-personalized VR-based system, where conventional cognitive tasks were operationalized in meaningful simulations of ADL's (Reh@City) and;
* a web tool which generates personalised paper and pencil tasks( Task Generator).

The investigators objective is to have a sample of 60 stroke patients between 40 and 70 years old, randomly allocated in three groups: the experimental group 1 were participants will perform 30 minutes of the VR training with Reh@City; the experimental group 2 were participants will perform 30 minutes of the paper and pencil training with the Task Generator, and the control group were participants will perform 30 minutes of conventional therapy (occupational therapy).

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke with more than 6 months post-stroke
* cognitive deficit but with enough capacity to understand the task and follow instructions with a minimum score of 11 over 17 in the Token Test (6-item version, Portuguese population)
* able to read and write

Exclusion Criteria:

* Neglect
* Severe depressive symptoms as assessed by the Beck Depression Inventory

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Montreal Cognitive Assessment | Baseline, End (4-6 weeks) and 8-weeks follow-up

SECONDARY OUTCOMES:
Change from baseline in the Trail Making Test A and B | Baseline, End (4-6 weeks) and 8-weeks follow-up
Change from baseline in the Verbal Paired Associates (WMS III) | Baseline, End (4-6 weeks) and 8-weeks follow-up
Change from baseline in the Digit Span (WAIS III) | Baseline, End (4-6 weeks) and 8-weeks follow-up
Change from baseline in the Symbol Search and Coding (WAIS III) | Baseline, End (4-6 weeks) and 8-weeks follow-up

OTHER OUTCOMES:
Crystallised Intelligence as assesed by Comprehension from the WAIS III | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Bermudez i Badia, PhD, Principal Investigator — Universidade da Madeira
Locations (1):
- Serviço de Saúde da Região Autónoma da Madeira, Funchal, Madeira, Portugal

REFERENCES:
- [Background] Faria, A. L., & Bermúdez i Badia, S. (2015). Development and evaluation of a web-based cognitive task generator for personalized cognitive training: a proof of concept study with stroke patients. In REHAB 2015: 3rd Workshop on ICTs for improving Patients Research Techniques. ACM.
- [Background] Faria, A. L., Vourvopoulos, A., Cameirão, M. S., Fernandes, J. C., & Bermúdez i Badia, S. (2014). An integrative virtual reality cognitive-motor intervention approach in stroke rehabilitation: a pilot study. In 10th ICDVRAT, Gothenburg, Sweden, Sept. 2-4, 2014.
- [Background] Vourvopoulos, A., Faria, A. L., Ponnam, K., & Bermúdez i Badia, S. (2014). RehabCity: Design and Validation of a Cognitive Assessment and Rehabilitation Tool through Gamified Simulations of Activities of Daily Living. In 11th International Conference on Advances in Computer Entertainment Technology. Funchal, Portugal.
- [Derived] Faria AL, Pinho MS, Bermudez I Badia S. A comparison of two personalization and adaptive cognitive rehabilitation approaches: a randomized controlled trial with chronic stroke patients. J Neuroeng Rehabil. 2020 Jun 16;17(1):78. doi: 10.1186/s12984-020-00691-5. PMID 32546251
- See also: Task Generator — http://neurorehabilitation.m-iti.org/TaskGenerator/